CLINICAL TRIAL: NCT00227617
Title: A Pilot Study of FOLFOX in Combination With Bevacizumab in Patients With Advanced Neuroendocrine Tumors
Brief Title: Combination Chemotherapy and Bevacizumab in Treating Patients With Advanced Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04458; NCI-2011-01214 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2019-12

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Lung Cancer; Neoplastic Syndrome; Neuroendocrine Tumor
Keywords: recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; pulmonary carcinoid tumor; gastrinoma; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma; recurrent islet cell carcinoma; metastatic gastrointestinal carcinoid tumor
MeSH Terms: conditions — Adenoma, Islet Cell; Lung Neoplasms; Neoplasms; Neuroendocrine Tumors; Gastrinoma; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma; Carcinoma, Islet Cell | interventions — Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FOLFOX with Bevacizumab (Experimental): Starting on Day 1, administered every two weeks:
  5-fluorouracil: 2400 mg/ m2 CIV; over 46-48 hours Leucovorin: 200 mg/ m2; over 2 hours Oxaliplatin : 85 mg/m2; over 2 hours Bevacizumab: 5 mg/kg IV over 30-90 minutes
  Interventions: Biological: bevacizumab; Drug: 5-fluorouracil; Drug: leucovorin; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — 5mg/kg IV q 2 wk on day 1. Initial study drug dose will be delivered over 90 +/- 15 minutes x1. If the first infusion is tolerated without fever/chills, the second infusion may be delivered over 60 +/- 10 minutes. If 60 minutes infusion is well tolerated, all subsequent infusions maybe be delivered over 30 +/- 10 minutes.
  Other Names: Avastin
Drug: 5-fluorouracil — 2400mg/m2 CIV over 46-48 hours D1-2 q2 weeks.
  Other Names: 5-FU; Adrucil
Drug: leucovorin — 200mg/m2 IV q2 wk on day 1 over a 2-hour period.
  Other Names: Folinic acid
Drug: oxaliplatin — 200mg/m2 IV q 2 wk on day 1 over a 2-hour period
  Other Names: Eloxatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of neuroendocrine tumors by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving combination chemotherapy together with bevacizumab and to see how well it works in treating patients with advanced neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of fluorouracil, leucovorin calcium, and oxaliplatin (FOLFOX) with bevacizumab in patients with advanced neuroendocrine tumors.
* Determine the best overall response rate in patients treated with this regimen.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the time to treatment failure and progression in patients treated with this regimen.
* Determine the biochemical marker response in patients treated with this regimen.

OUTLINE: This is an open-label, pilot study. Patients are stratified according to tumor type (carcinoid vs islet cell vs poorly differentiated neuroendocrine).

Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46-48 hours beginning on day 1. Patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 14 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 39-102 patients (13-34 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed neuroendocrine tumor (NET)

  * Carcinoid at any site, with or without carcinoid syndrome
  * Pancreatic islet cell tumor

    * Prior streptozocin-based therapy not required
  * Poorly differentiated NET of any primary site (this arm closed to accrual May 2009)

    * Progression with prior treatment with cisplatin-, or carboplatin-based chemotherapy required (unless contraindicated)
* The following tumors are not allowed:

  * Endocrine organ carcinoma
  * Adrenal gland malignancies
  * Thyroid carcinoma of any histology
  * Pheochromocytoma/paraganglioma
* Advanced disease

  * Disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
* Radiologically or clinically confirmed progressive disease

  * At least 25% increase in radiologically or clinically measurable disease
  * At least 20% increase in the longest diameter (LD) of any previously documented lesion
  * Increase in the sum of the LD of multiple lesions in aggregate of 20%, OR appearance of new lesions OR deterioration in clinical status
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional radiographic techniques OR ≥ 10 mm by spiral CT scan

    * Ultrasound or positron-emission tomography alone not sufficient
  * Bone lesions, ascites, peritoneal carcinomatosis, pleural or pericardial effusion, and irradiated lesions are not considered measurable disease
* Primary tumors of the pancreas should not invade adjacent organs (e.g., stomach or duodenum)
* No history or evidence of brain or leptomeningeal disease (baseline CNS imaging required if clinical suspicion of CNS metastases)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No history of hemoptysis or bleeding diathesis
* No coagulopathy unrelated to therapeutic anticoagulation
* No significant bleeding events within the past 6 months unless the source of the bleeding has been resected

Hepatic

* Bilirubin < 2 mg/dL
* ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if due to liver metastases)

Renal

* Creatinine ≤ 2 mg/dL
* Protein ≤ 1+ OR
* Protein < 1 gm on 24-hour urine collection
* Urine protein:creatinine ratio < 1.0

Cardiovascular

* History of thromboembolic condition allowed provided patient is on therapeutic anticoagulation at a stable dose for ≥ 4 weeks

  * Concurrent daily prophylactic aspirin (< 325 mg/day) allowed
* No uncontrolled hypertension, myocardial infarction, clinically significant peripheral arterial ischemia, visceral arterial ischemia or angina within the past 6 months
* No serious cardiac arrhythmia requiring medication
* No cerebrovascular event (e.g., stroke or transient ischemic attack) within the past 12 months
* No history of peripheral vascular disease ≥ grade 2
* No history New York Heart Association class II-IV congestive heart failure
* Blood pressure ≤ 160/90 mm Hg

Gastrointestinal

* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No predisposing uncontrolled small bowel or colonic disorder

  * Baseline disease-related diarrhea allowed if symptoms are stable and well-characterized (i.e., # stools/day stable)
* No gastric or esophageal varices
* No gastroduodenal ulcers determined to be active by endoscopy

Pulmonary

* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis
* No lung tumor in close proximity to a major vessel, or with associated cavitation
* No pleural effusion or ascites that causes ≥ grade 2 dyspnea

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after completion of study treatment
* No significant traumatic injury within the past 28 days
* No currently active second malignancy other than, non-melanoma skin cancer or carcinoma in situ

  * Patients are not considered to have a currently active malignancy if they have completed therapy and are considered by their physician to be at ≤ 30% risk for relapse
* No known hypersensitivity reaction attributed to study drugs or to compounds of similar chemical or biological composition
* No symptomatic peripheral neuropathy > grade 1
* No other severe disease or comorbidity that would preclude study participation
* No medically uncontrolled seizures
* No active infection
* No serious non-healing wound, ulcer, or bone fracture
* No psychiatric illness or social situation that would preclude study compliance
* No other severe, concurrent disease, infection, or co-morbidity that in the judgement of the investigator would constitute a hazard for study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior cytokine therapy
* At least 4 weeks since prior immunotherapy
* No prior tyrosine kinase inhibitors or anti-vascular endothelial growth factor (VEGF) angiogenic inhibitors

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No prior oxaliplatin
* Prior chemoembolization therapy allowed provided it did not affect areas of measurable disease

Endocrine therapy

* Prior and concurrent somatostatin analogs allowed for symptomatic control and/or control of hormone hypersecretion only provided treatment was initiated > 3 months prior to study entry

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

  * Prior radiotherapy must not affect areas of measurable disease
* No concurrent radiotherapy to only site of measurable disease

Surgery

* Recovered from prior surgery
* Prior cryotherapy allowed provided it did not affect areas of measurable disease
* At least 28 days since prior major surgical procedure or open biopsy
* At least 7 days since minor surgical procedure, fine-needle aspirations, or core biopsy
* No prior organ allograft
* No concurrent major surgery

Other

* At least 4 weeks since prior participation in an experimental drug study
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No halogenated antiviral agents
* Concurrent antiplatelet agents allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06-08 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Bergsland, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Univeristy of California, San Francisco, San Francisco, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Simon 2-stage design: 13 patients in stage 1. If at least 2 objective tumor responses were observed by 12 cycles of therapy, the cohort was to be expanded to enroll a total of 39 treated patients.
Groups:
- Carcinoid; PNET; Poorly Differentiated Neuroendocrine Carcinomas (PDNEC): Starting on Day 1, administered every two weeks:
  * Leucovorin: 200 mg/ m2; over 2 hours
  * Oxaliplatin : 85 mg/m2; over 2 hours
  * followed by 5-fluorouracil (5-FU): 2400 mg/ m2 CIV; over 46-48 hours
  * Bevacizumab: 5 mg/kg IV
    5-FU bolus was permanently dropped after nearly all of the first 13 patients required a dose reduction for toxicity:
  * 3 in carcinoid
  * 10 in PNET
Period: Stage 1
Arm/Group | Carcinoid | PNET | Poorly Differentiated Neuroendocrine Carcinomas (PDNEC)
Started | 22 | 12 | 2
Completed | 22 | 12 | 2
Not Completed | 0 | 0 | 0
Period: Stage 2
Arm/Group | Carcinoid | PNET | Poorly Differentiated Neuroendocrine Carcinomas (PDNEC)
Started (Study was terminated due to low accrual) | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient data was migrated at time of close to accrual and the treatment arm information was not included in data migration. As such baseline data for patients with Carcinoid Neuroendocrine Tumors, Pancreatic Neuroendocrine Tumors, Poorly Differentiated Neuroendocrine Carcinoma data has been reported across treatment arms
Groups:
- Combined Neuroendocrine Tumors: Patients with Carcinoid Neuroendocrine Tumors, Pancreatic Neuroendocrine Tumors, and Poorly Differentiated Neuroendocrine Carcinoma enrolled on the protocol
Arm/Group | Combined Neuroendocrine Tumors
Number analyzed (Participants) | 36
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 6
  50-59 years old | 13
  60-69 years old | 13
  70-79 years old | 3
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 28
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Discontinuation Due to Adverse Events Possibly Related to Study Treatment
Description: Rates of discontinuation were calculated as counts and percentages of patients whom discontinued treatment due to adverse events possibly related to the investigational treatments not including neuropathy.
Time Frame: From beginning of treatment up to 18 months; Post-study survival follow-up up to 8 years
Population: Study terminated early due to low accrual. UCSF moved its clinical research database from Velos to OnCore in July 2010 and some of the data for this study was not transferred. Results reported accurate to date
Measure: Count of Participants; unit: Participants
Groups:
- Carcinoid; PNET; PDNEC: Starting on Day 1, administered every two weeks:
  5-fluorouracil: 2400 mg/ m2 CIV; over 46-48 hours Leucovorin: 200 mg/ m2; over 2 hours Oxaliplatin : 85 mg/m2; over 2 hours Bevacizumab: 5 mg/kg IV over 30-90 minutes
  bevacizumab: 5mg/kg IV q 2 wk on day 1. Initial study drug dose will be delivered over 90 +/- 15 minutes x1. If the first infusion is tolerated without fever/chills, the second infusion may be delivered over 60 +/- 10 minutes. If 60 minutes infusion is well tolerated, all subsequent infusions maybe be delivered over 30 +/- 10 minutes.
  5-fluorouracil: 2400mg/m2 CIV over 46-48 hours D1-2 q2 weeks.
  leucovorin: 200mg/m2 IV q2 wk on day 1 over a 2-hour period.
  oxaliplatin: 200mg/m2 IV q 2 wk on day 1 over a 2-hour period
Arm/Group | Carcinoid | PNET | PDNEC
Number analyzed (Participants) | 22 | 12 | 2
Participants | 3 | 3 | 0

2. Primary Outcome: Best Objective Response
Description: Best Objective Response by RECIST with Exact 95% Binomial CIs across all tumor types. The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria Target lesions response + Non-Target lesions response + Evaluation of non-target lesions (Yes / No) = Overall response
Time Frame: From Baseline until disease progression, up to 8 years
Population: Intent-to-Treat population used for analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Combined Neuroendocrine Tumors: Patients with Carcinoid Neuroendocrine Tumors, Pancreatic Neuroendocrine Tumors, Poorly Differentiated Neuroendocrine Carcinoma who received at least one treatment
Arm/Group | Combined Neuroendocrine Tumors
Number analyzed (Participants) | 36
percentage of participants
  Unevaluable | 2.8 [0 to 14]
  Progressive Disease | 2.8 [0 to 14]
  Partial Response | 31 [16 to 48]
  Stable Disease | 64 [46 to 79]

3. Secondary Outcome: Time to Progression
Description: Time to disease progression will be defined as the time from baseline until documented disease progression or death (whichever occurs first).
Time Frame: From beginning of treatment up to 18 months; Post-study survival follow-up up to 8 years
Population: A reliable median and 95% confidence interval for time to progression could not be computed for participants with Poorly Differentiated Neuroendocrine Carcinoma (PDNEC) due to the insufficient number of participants with this condition (N=2)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carcinoid: Carcinoid Neuroendocrine Tumors
- PNET: Pancreatic Neuroendocrine Tumors
- PDNEC: Poorly Differentiated Neuroendocrine carcinoma
Arm/Group | Carcinoid | PNET | PDNEC
Number analyzed (Participants) | 22 | 12 | 0
months | 19.3 [9.9 to 29.9] | 21 [7.4 to 31.4] |

4. Secondary Outcome: Overall Median Survival
Description: The overall survival is defined as the time from baseline until death (Carcinoid, PNET, PDNEC) using Kaplan-Meier Survival analysis methods.
Time Frame: until death, up to 8 years
Population: Intent-to-Treat population used for analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Neuroendocrine Tumors
Number analyzed (Participants) | 36
months | 31.0 [23.3 to 34.5]

5. Secondary Outcome: Overall Time to Treatment Failure
Description: Time to treatment failure is defined as the time from the initial complete or partial response to documented disease progression or death (whichever occurs first) across treatment groups and inclusive of drug holidays and estimated using Kaplan-Meier survival analysis methods
Time Frame: From initial complete or partial response to disease progression, up to 8 years
Population: Intent-to-Treat population used for analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combined Neuroendocrine Tumors
Number analyzed (Participants) | 36
months | 9.1 [6.5 to 13.8]

6. Secondary Outcome: Biochemical Marker Response
Description: Biochemical marker response is defined as >=50% reduction in marker or hormone(s) that were elevated at baseline. Markers/hormones tested are: Chromagranin A (CGA), 5-HIAA, Insulin, Proinsulin, C-peptide, Pancreatic polypeptide, Gastrin, Glucagon, and Vasointestinal Peptide.
Time Frame: From Baseline until end of treatment, up to 8 years
Population: Percentages of participants who met criteria of a biochemical marker response are also displayed
Measure: Number; unit: percentage of participants
Groups:
- PDNEC: Poorly differentiated neuroendocrine carcinoma (PDNEC)
Arm/Group | Carcinoid | PNET | PDNEC | All Neuroendocrine Tumors
Number analyzed (Participants) | 13 | 10 | 2 | 23
percentage of participants
  Chromogranin A (CGA) | 25 | 78 | 0 | 50
  Any hormone and/or CGA | 31 | 80 | 0 | 52
  Any hormone (not including CGA): number analyzed (Participants) | 13 | 5 | 2 | 18
  Any hormone (not including CGA) | 23 | 60 | 0 | 33

ADVERSE EVENTS:
Time Frame: Up to 8 years
Description: Data migration issue prevented this data from being reported by treatment arm. Adverse Events grade 3 and higher were not reported.
Groups:
- Combined Neuroendocrine Tumors: Patients enrolled on protocol with Carcinoid Neuroendocrine Tumors, Pancreatic Neuroendocrine Tumors, or Poorly Differentiated Neuroendocrine Carcinoma whom received at least one treatment
Arm/Group | Combined Neuroendocrine Tumors
All-Cause Mortality (participants affected / at risk) | 3/36
Serious Adverse Events (participants affected / at risk) | 12/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Neuroendocrine Tumors (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Constitutional Symptoms (General disorders) | 1
Fatigue (General disorders) | 1 — asthenia, lethargy, malaise
Fever (General disorders) | 1 — in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Perforation, GI - Small bowel NOS (Gastrointestinal disorders) | 2
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 1
Hemorrhage, GI- Upper GI NOS (Gastrointestinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 1 — (fever of unknown origin without clinically or microbiologically documented infection) (AND<1.0 X 10e9/L, fever >38.5 degrees)
Infection - Other (specify,__) (Infections and infestations) | 2
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 3
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Neuroendocrine Tumors (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 8 (31)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (40)
Platelets (Blood and lymphatic system disorders) | 8 (29)
Other (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 8 (15)
Fatigue (General disorders) | 32 (78)
Weight Loss (Gastrointestinal disorders) | 10 (13)
Anorexia (Gastrointestinal disorders) | 17 (25)
Constipation (Gastrointestinal disorders) | 19 (30)
Diarrhea (Gastrointestinal disorders) | 26 (56)
Mucositis/stomatitis (Gastrointestinal disorders) | 3 (6)
Perforation, GI - Small bowel NOS (Gastrointestinal disorders) | 2 (2)
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 (1)
Febrile Neurtropenia (Blood and lymphatic system disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 9 (27)
Neuropathy: sensory (Nervous system disorders) | 34 (144)
Pain- Abdominal (Gastrointestinal disorders) | 15 (34)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Technical problems with database migration lead to missing treatment assignment values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes